CLINICAL TRIAL: NCT02099305
Title: Impact of Increasing Adolescent Depression Literacy on Treatment-Seeking Behavior
Brief Title: Randomized, School-based Effectiveness Trial of the Adolescent Depression Awareness Program
Acronym: ADAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Holly C. wilcox, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1-wilcox; R01MH095855 (NIH)
Record Dates: First submitted 2014-03-20; First posted 2014-03-28 (Estimated); Last update posted 2017-06-12 (Actual); Status verified 2016-03

CONDITIONS: Adolescent - Emotional Problem; Depression; Prevention Harmful Effects
Keywords: Adolescent; Depression; Early intervention (education); Randomized Controlled Trial; Primary Prevention; schools; Health Literacy; Discrimination (Psychology); Mental Health Services
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Receive Adolescent Depression Awareness Program (ADAP) intervention
  Interventions: Other: Adolescent Depression Awareness Program (ADAP)
- Wait list control (No Intervention): no intervention

INTERVENTIONS:
Other: Adolescent Depression Awareness Program (ADAP) — Depression education curriculum delivered by trained school health education teachers or other school personnel
  Other Names: ADAP
  Arms: Intervention

SUMMARY:
The primary goal of the proposed research is to assess the effectiveness of the Adolescent Depression Awareness Program (ADAP), a school-based depression education program, in increasing depression literacy and treatment seeking in high school students. The ADAP intervention will be carried out in approximately 60 schools with over 15,000 students. The following are ADAP Implementation Sites: Baltimore Archdiocese High Schools; New Castle County, Delaware; Washtenaw County, Michigan; and York County, Pennsylvania.

DETAILED DESCRIPTION:
The primary goal of the proposed research is to assess the effectiveness of the Adolescent Depression Awareness Program (ADAP), a school-based depression education program, in increasing depression literacy and treatment seeking. This proposal will have broad reach as the intervention will be carried out in 66 schools with over 15,000 students.

The lifetime prevalence of Major Depressive Disorder (MDD) in the United States is high, ranging from 15% to 17%. Its usual symptom onset occurs early in life, during teen or young adult years. It has been estimated that 8.5% of youth ages 12 to 17 (over 2 million adolescents) experienced at least one Major Depressive Episode in the past year (SAMHSA Office of Applied Studies, 2008). Nearly half (48.3%) of these youth reported severe impairment in at least one of four major role domains (home, school/work, family relationships, or social life). The onset of depression during adolescence is associated with increased risks for educational underachievement, unemployment, early parenthood, substance dependence, anxiety disorders, and recurrent major depression during early adulthood (Fergusson & Woodward, 2002). The most severe consequence of untreated depression is suicide. Psychological autopsy studies of adolescent suicides have reported that upwards of 90% had at least one psychiatric disorder at the time of their death, most notably depression (Marttunen et al., 1990; Brent et al., 1993; Shaffer et al., 1996). From a developmental perspective, the prevention and treatment of depression during adolescence can provide lifelong benefits. Effective treatments for adolescent depression are available (TADS, 2007); however, adolescents in need of treatment are often not recognized by parents, teachers, or peers. The National Comorbidity Study-Replication estimated a median delay of 8 years between the onset of depressive symptoms and receiving treatment (Wang et al., 2006). The early identification of depression leading to effective treatment can help address the morbidity and mortality associated with adolescent depression.

Despite the importance of adolescent depression, there have been few large-scale randomized trials investigating the effectiveness of universal interventions targeting depression among adolescents. ADAP is a 3-hour high school-based curriculum, proposed herein to be delivered as part of the standard high school health education curriculum, aimed at improving depression literacy. The mission of ADAP is to educate high school students, teachers, and parents about teenage unipolar and bipolar depression (Hess et al., 2004). The core message of ADAP is that "depression is a treatable medical illness." ADAP was developed in 1999 by a team of psychiatrists and psychiatric nurses from the Johns Hopkins University School of Medicine. In the past decade, ADAP has been implemented in over 85 schools with over 20,000 students throughout the United States. Previously published research evaluating ADAP described a significant improvement in adolescents' knowledge about depression after receiving the curriculum using a one group pretest/posttest design (Swartz et al., 2008). Recently, in Tulsa, Oklahoma, comparison schools were included, and it was found that the proportion of students achieving "depression literacy" (scoring 80% or higher on our knowledge assessment) more than tripled from pretest to posttest (Leon et al., in review) in the ADAP group. To date, a randomized design has not been employed and the impact of ADAP on treatment seeking behaviors has not been studied. Both of these issues are important to address before ADAP can be routinely integrated into high school health education curricula. The specific aims of this proposal are as follows:

Specific Aim 1: To assess the effectiveness of ADAP, a school-based depression education program, in increasing depression literacy.

1.1 To assess depression literacy changes following the intervention, as compared to the standard health education curriculum, with a post-test at 6 weeks post intervention.

1.2 To assess the sustainability of depression literacy changes with a post-test at 4 months post ADAP.

Specific Aim 2: To assess whether the ADAP intervention, as compared to the standard health curriculum, has an influence on treatment seeking behaviors in high school students, as measured by an increase in visits to school counselors and self-reported treatment seeking.

2.1 To track mental health help-seeking and the receipt of mental health services pre and post ADAP in a subset of schools (28 schools in York County Pennsylvania and St. Francis Indian School on the Rosebud Indian Reservation served by the Indian Health Service).

2.2 To track mental health visits to school counselors in aggregate pre and post ADAP in all 66 participating schools.

Specific Aim 3: To identify possible mediators (e.g., fidelity) and moderators of intervention impact (e.g., access to community mental health services, teacher characteristics, school characteristics, parental participation in the community forum; stigma).

ELIGIBILITY:
Inclusion Criteria:

* enrolled in one of the participating schools parental consent and student assent is required for the web-based survey

Exclusion Criteria:

* not enrolled in the participating schools

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17000 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Adolescent Depression Knowledge Questionnaire (ADKQ) | Change from pretest (directly before intervention) to post-test (6 weeks after ADAP). We will see if this is sustained 4 months after ADAP.
  The Adolescent Depression Knowledge Questionnaire (ADKQ) will be used to assess depression literacy

SECONDARY OUTCOMES:
Reported and Intended Behaviour Scale (RIBS) | Change from pretest (directly before intervention) to post-test (6 weeks after ADAP). We will see if this is sustained 4 months after ADAP.
  The Reported and Intended Behaviour Scale (RIBS) will be used to assess mental health stigma.

OTHER OUTCOMES:
Help-seeking and the receipt of Mental Health Services | after the ADAP intervention
  We have designed a web-based survey in RedCAP to assess help-seeking and the receipt of Mental Health Services, barriers and attitudes, and other issues among students in York County, Pennsylvania with parental consent.

CONTACTS AND LOCATIONS:
Overall Officials: Holly C. Wilcox, PhD, Principal Investigator — Associate Professor, Johns Hopkins School of Medicine; Karen Swartz, MD, Study Chair — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Johns Hopkins, Baltimore, Maryland

REFERENCES:
- [Result] Ruble AE, Leon PJ, Gilley-Hensley L, Hess SG, Swartz KL. Depression knowledge in high school students: effectiveness of the adolescent depression awareness program. J Affect Disord. 2013 Sep 25;150(3):1025-30. doi: 10.1016/j.jad.2013.05.033. Epub 2013 Jun 18. PMID 23790814
- [Result] Swartz KL, Kastelic EA, Hess SG, Cox TS, Gonzales LC, Mink SP, DePaulo JR Jr. The effectiveness of a school-based adolescent depression education program. Health Educ Behav. 2010 Feb;37(1):11-22. doi: 10.1177/1090198107303313. Epub 2007 Jul 25. PMID 17652614
- [Result] Hess SG, Cox TS, Gonzales LC, Kastelic EA, Mink SP, Rose LE, Swartz KL. A survey of adolescents' knowledge about depression. Arch Psychiatr Nurs. 2004 Dec;18(6):228-34. doi: 10.1016/j.apnu.2004.09.005. PMID 15625662
- [Derived] Townsend L, Musci R, Stuart E, Heley K, Beaudry MB, Schweizer B, Ruble A, Swartz K, Wilcox H. Gender Differences in Depression Literacy and Stigma After a Randomized Controlled Evaluation of a Universal Depression Education Program. J Adolesc Health. 2019 Apr;64(4):472-477. doi: 10.1016/j.jadohealth.2018.10.298. Epub 2019 Jan 4. PMID 30612807
- [Derived] Swartz K, Musci RJ, Beaudry MB, Heley K, Miller L, Alfes C, Townsend L, Thornicroft G, Wilcox HC. School-Based Curriculum to Improve Depression Literacy Among US Secondary School Students: A Randomized Effectiveness Trial. Am J Public Health. 2017 Dec;107(12):1970-1976. doi: 10.2105/AJPH.2017.304088. Epub 2017 Oct 19. PMID 29048969
- See also: Adolescent Depression Awareness Program (ADAP) website — http://www.hopkinsmedicine.org/psychiatry/specialty_areas/moods/ADAP/